CLINICAL TRIAL: NCT02249507
Title: Aerobic Exercise in Postexercise Cardiovascular Responses in Resistant Hypertension: a Cross-over Randomized Controlled Trial
Brief Title: Aerobic Exercise in Postexercise Cardiovascular Responses in Resistant Hypertension: a Cross-over Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 13-0309; 13-0309 (Other: CEP-HCPA)
Record Dates: First submitted 2014-09-23; First posted 2014-09-25 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-08

CONDITIONS: Hypertension
Keywords: Resistant Hypertension; Aerobic Exercise
MeSH Terms: conditions — Hypertension | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (No Intervention): sited rest for 45 minutes
- higher intensity aerobic exercise (Experimental): 45 minutes of aerobic exercise at 75%HRmax
  Interventions: Other: aerobic exercise
- lower intensity aerobic exercise (Experimental): 45 minutes of aerobic exercise at 50%HRmax
  Interventions: Other: aerobic exercise

INTERVENTIONS:
Other: aerobic exercise — aerobic exercise (cycloergometer) at selected intensity (HRmax or equivalent)
  Arms: higher intensity aerobic exercise; lower intensity aerobic exercise

SUMMARY:
Aerobic exercise has the potential to diminish blood pressure values. The aim of this study is to determine whether this potential is also applicable for those with resistant hypertension and whether exercise intensity plays a role in this context. We hypothesize that performing an aerobic exercise session reduces blood pressure values in resistant hypertensive patients in a dose-response relation with exercise intensity.

DETAILED DESCRIPTION:
Exercise prescription is gathering great importance in preventive health. Several organizations endorse the performance of at least 150min/wk of moderate intensity or 75min/wk of higher intensities in order to achieve better health parameters in different contexts. Aerobic exercise is known to be an effective way to diminish BP levels post-session. These responses are widely applicable in hypertensive subjects, acting in aid of BP management treatment. Although these benefits of aerobic exercise are well known, few studies explore the potential of this intervention in resistant-to-treatment patients. Moreover, the effects different intensities of aerobic exercise in this population is scarce. Thus, the aim of this study is to determine the magnitude of BP responses, if there is any, of resistant hypertensive subjects to two different intensities of aerobic exercise, compared with a control session. For that, subjects will be enrolled for one pre-intervention cardiopulmonary exercise testing and three randomized intervention sessions: control, 50%HRmax and 75%HRmax. Prior and immediately after all intervention sessions (during 1h), forearm blood flow and reactive hyperemia will be assessed by venous occlusion plethysmography. After the sessions, 24h blood pressure will be assessed with an ambulatory blood pressure monitoring system.

ELIGIBILITY:
Inclusion Criteria:

resistant-to-treatment hypertensive subjects (24h ambulatory BP above 130/80, or daytime ambulatory BP above 135/85, or night-time ambulatory BP above 120/70 in spite use of 3 anti-hypertensive medications of different classes, being one diuretic; or use of 4 or more anti-hypertensive medications).

Exclusion Criteria:

Muscle or skeletal abnormalities that preclude effort, abnormal exercise stress test, major illnesses that would preclude exercise effort or could influence in the outcome variables (pulmonary disease, valve disease, renal insufficiency, etc.)

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2013-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Ambulatory Blood Pressure Monitoring | 22h

SECONDARY OUTCOMES:
Forearm blood flow | 1h
  Accessed by venous occlusion plethysmography. Compared with pre-intervention values
Reactive hyperemia | pre and 30min post
  Accessed by venous occlusion plethysmography.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Umpierre, PhD, Principal Investigator — Federal University of Health Science of Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil